CLINICAL TRIAL: NCT06618976
Title: SOTA-THROMBOSIS: Antithrombotic Activities of Sotagliflozin vs. Empagliflozin
Brief Title: Antithrombotic Activities of Sotagliflozin vs. Empagliflozin
Acronym: SOTATHROMBUS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Juan Badimon, Professor of Medicine, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-24-00304
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Thrombosis
Keywords: Thrombosis; Platelets; Heart failure; SGLT2; SGLT1/2
MeSH Terms: conditions — Thrombosis; Heart Failure | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; empagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sotagliflozin then Empagliflozin (Other): Subjects randomized to 'Arm A' will receive 1-month of 'Sotagliflozin' treatment first and then 1-month of 'Empagliflozin' treatment second, separated by a 1-month of washout period.
  Interventions: Drug: Sotagliflozin; Drug: Empagliflozin
- Empagliflozin then Sotagliflozin (Other): Subjects randomized to 'Arm B' will receive1-month of 'Empagliflozin' treatment first and then1-month of 'Sotagliflozin' treatment second, separated by a 1-month of washout peri od
  Interventions: Drug: Sotagliflozin; Drug: Empagliflozin

INTERVENTIONS:
Drug: Sotagliflozin — Sotagliflozin 400 mg, P.O. once daily for 1 month.
Drug: Empagliflozin — Empagliflozin 10 mg, P.O. once daily for 1 month.

SUMMARY:
The availability of Sodium-glucose cotransporter-2 inhibitors (SGLT2-i) has dramatically altered the management of heart failure (HF) patients, independently of their ejection fraction and glycemic status. A meta-analysis of 57 studies comparing SGLT2-I monotherapy vs. placebo or active comparator showed reductions in major cardiovascular events, but no impact on atherothrombotic events. In fact, a non-significant increase in the risk for non-fatal stroke was observed. Similar trend observed in multiple trials indicate a SGLT2-i class effect. Sotagliflozin is the first dual SGLT1/2 receptor inhibitor, that was shown to significantly reduce atherothrombotic events compared with placebo in diabetic HF patients, suggesting that dual SGLT1/2 inhibitor may have additional properties vs. SGLT2-i. The hypothesis of this study is that dual SGLT1/2 inhibition by sotagliflozin improves thrombogenic profile (i.e. reduces thrombus formation), which could make it a safer and more effective treatment option for cardiovascular (CV) patients than SGLT2-i. To test the hypothesis, the researchers will compare the antithrombotic activity of sotagliflozin vs. empagliflozin in healthy volunteers using a randomized, cross-over study design, where each participant will receive both study treatments (sotagliflozin and empagliflozin) separated by a washout period. Treatment effects will be assessed by measuring ex vivo thrombus formation using the Badimon Perfusion chamber, platelet aggregation using Multiplate Analyzer, and Thromboelastometry using RoTEM Gamma. Study assessments will be performed before initiating (baseline/pre-treatment) and after completion of each treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible if they meet all of the following criteria:

* Male or female volunteers older than 18 years old.
* Disease-free as assessed by medical history and physical examination.
* Ability to provide signed informed consent.

Exclusion criteria:

Subjects will be excluded if they meet any of the following criteria:

* Pregnant or lactating women
* History of clinically relevant cardiovascular, pulmonary, hepatic, gastrointestinal, renal, metabolic, hematologic, neurologic, respiratory or psychiatric disease, bleeding, acute infectious disease or signs of acute illness.
* Use of medication within one month prior to study drug administration or within six times the elimination half-life (whichever is longer), except for oral contraceptives or occasional use of acetaminophen or an antihistamine.
* History of drug abuse or alcohol consumption >20 g/day [125 ml (30ml=1oz) glass of 10% wine = 12.5 g, 40 mL aperitif of 40% = 17 g, 250 mL glass of 6% beer = 15g]
* Loss of >400 mL blood or blood donation within 3 months.
* Conditions associated with hemorrhagic risk, e.g., frequent epistaxis, gastrointestinal ulcer, hemorrhagic vascular lesions, recent surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Thrombus size | Baseline and end of each treatment period (1 month and 3 months)
  Changes in blood thrombogenicity (thrombus size) from baseline to post-treatment

SECONDARY OUTCOMES:
Platelet aggregation | Baseline and end of each treatment period (1 month and 3 months)
  A platelet aggregation is a blood test that looks at the reactivity of platelets.
Clot formation size | Baseline and end of each treatment period (1 month and 3 months)
  The size of the clot will be assessed in whole blood samples using a thromboelastometry

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Badimon, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Requena-Ibanez JA, Zafar MU, Ferrandez-Escarabajal M, Escolar G, Santos-Gallego C, Lam D, Badimon JJ. Rationale and Design of the SOTA-THROMBOSIS Trial (ATRU-VI): Antithrombotic Activities of Sotagliflozin Compared With Empagliflozin. J Cardiovasc Pharmacol. 2025 Nov 1;86(5):458-462. doi: 10.1097/FJC.0000000000001747. PMID 40748666